CLINICAL TRIAL: NCT00554268
Title: An Open Label Phase I Trial of PBI-05204 in Advanced Cancer Patients
Brief Title: Trial of PBI-05204 in Advanced Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0375
Record Dates: First submitted 2007-11-02; First posted 2007-11-06 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2013-04

CONDITIONS: Solid Tumors
Keywords: Advanced Cancers; Solid Tumors; PBI-05204
MeSH Terms: interventions — PBI-05204

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PBI-05204 (Experimental): PBI-05204 starting dose = 0.0083 mg/kg/day by mouth (PO) x 3 weeks per cycle.
  Interventions: Drug: PBI-05204

INTERVENTIONS:
Drug: PBI-05204 — Starting dose = 0.0083 mg/kg/day by mouth (PO) x 3 weeks per cycle

SUMMARY:
The goal of this clinical research study is to find the highest safe dose of PBI-05204 that can be given to patients with advanced solid tumors. The study will also look at how PBI-05204 is processed by the body, how it leaves the body, how it affects the body, and if it is affecting certain proteins in the cancer cells.

DETAILED DESCRIPTION:
The Study Drug PBI-05204, made from the oleander plant, is designed to prevent the growth of cancer cells by affecting proteins that lead to cell death.

Screening Tests

Before you can begin receiving the study drug, you will have "screening tests" to help the doctor decide if you are eligible to take part in this study. The following tests will be performed:

* You will have a physical exam, including measurement of vital signs (blood pressure, heart rate, temperature, and breathing rate), height, and weight.
* You will be asked how well you are able to perform the normal activities of daily living (performance status evaluation).
* Your complete medical history will be recorded.
* You will have an electrocardiogram (ECG -- a test that measures the electrical activity of the heart).
* You may have an echocardiogram (a picture of your heart using sound waves), if applicable.
* You will have a computed tomography (CT) scan or magnetic resonance imaging (MRI) to check the status of the disease.
* Blood (about 3-4 teaspoons) and urine will be collected for routine tests.
* Women who are able to have children must have a negative blood (about 2 teaspoons) or urine pregnancy test.

Study Drug Dose Level:

If you are found to be eligible to take part in this study, the amount of PBI-05204 that you take will be based on how many participants have been enrolled before you, and on the safety information that is available. There may be up to 6 participants enrolled in each group. The first group of participants enrolled on this study will receive PBI-05204 at the lowest dose level. If no intolerable side effects are experienced, the next group of participants will take a higher dose level. This process will continue until researchers find the highest dose of PBI-05204 that can be given without intolerable side effects occurring.

Study Drug Administration:

Depending on which group you are enrolled in, you will take the PBI-05204 capsules by mouth every day at the same time or twice a day (every 12 hours). Your Doctor will tell you which schedule you are on. You will take the drug on Days 1-21. On Days 22-28 you will take no study drug. Each 28 days is called a "study cycle".

Study Visits:

At the Predose Visit, 1-7 days before Day 1 of Cycle 1 you will have the following tests and procedures performed:

* You will have a physical exam, including measurement of your vital signs, height, and weight.
* You will have a performance status evaluation.
* Urine will be collected for routine tests.
* You will have an ECG, if applicable
* You will have your heart rate monitored by a Holter monitor. A Holter monitor is a machine that continuously records the heart's rhythms. Electrodes (small conducting patches) are stuck onto your chest and attached to a small recording monitor. You carry the Holter monitor in a pocket or in a small pouch worn around your neck or waist. The monitor is battery operated. After 24 hours, you return the monitor to the study doctor. The study doctor will look at the records and see if there have been any irregular heart rhythms.
* Blood (about 3-4 teaspoons) will be collected for routine tests.
* Women who are able to have children will have a blood (about 2 teaspoons) or urine pregnancy test.

On Day 1 Cycle 1 you will have the following tests and procedures performed:

* You will have a physical exam, including measurement of your vital signs.
* You will have a performance status evaluation.
* You will have an ECG. The ECG will be repeated on Day 1 of every later Cycle.
* Blood (about 3-4 teaspoons) and urine will be collected for routine tests.
* You will take your dose of PBI-05204 by mouth.
* Blood (about 2 teaspoons each time) will be collected for PK testing before you take the first daily dose of the study drug and then 1, 2, 4, 6, and 8 hours later.
* Blood (about 6 teaspoons) will be collected for pharmacodynamic (PD) testing before you take the study drug. PD testing is used to look at how the level of study drug in your body may affect the disease.

On Day 2 of Cycle 1 you will have the following:

* You will take your dose of PBI-05204 by mouth
* You will have an ECG.

On Day 7 of Cycle 1 you will have the following:

* Blood (about 6 teaspoons) will be drawn for PD testing.
* You will take your dose of PBI-05204 by mouth.
* You will have your heart rate monitored by a Holter monitor.

On Day 8 of Cycle 1 you will have the following tests and procedures performed:

* You will have a physical exam, including measurement of your vital signs.
* You will have a performance status evaluation.
* Blood (about 3-4 teaspoons) and urine will be collected for routine tests.
* You will take your dose of PBI-05204 by mouth.
* Blood (about 2 teaspoons each time) will be collected for PK testing before you take the first daily dose of the study drug and then 1, 2, 4, 6, and 8 hours later. Additional blood (about 2 teaspoons each time) will also be collected for PK testing before you take the second daily dose of the study drug and then 1, 2, 4, and 12 hours later.
* You will have an ECG.

On Day 15 of Cycle 1 you will have the following tests and procedures performed:

* You will have a physical exam, including measurement of your vital signs.
* You will have a performance status evaluation.
* You will have an ECG.
* Blood (about 3-4 teaspoons) and urine will be collected for routine tests.
* You will take your dose of PBI-05204 by mouth.
* Blood (about 2 teaspoons each time) will be collected for PK testing before you take the first daily dose of the study drug and then 1, 2, 4, 6, and 8 hours later.

On Day 21 of Cycle 1 you will have the following tests and procedures performed:

* You will have a physical exam, including measurement of your vital signs.
* You will have a performance status evaluation.
* Blood (about 3-4 teaspoons) and urine will be collected for routine tests.
* You will take your dose of PBI-05204 by mouth.
* Blood (about 2 teaspoons each time) will be collected for PK testing before you take the first daily dose of the study drug and then 1, 2, 4, 6, and 8 hours later. Additional blood (about 2 teaspoons each time) will also be collected for PK testing before you take the second daily dose of the study drug and then 1, 2, 4, and 12 hours later.
* Blood (about 6 teaspoons) will be collected for PD testing.

During the last week of Cycle 2, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs, height and weight.
* You will have a performance status evaluation.
* Blood (about 3-4 teaspoons) and urine will be collected for routine tests.
* You will have a CT or MRI scan to check the status of the disease.
* Women who are able to have children will have a blood (about 2 teaspoons) or urine pregnancy test.

On Day 1 of Cycles 3 and beyond you will have a physical exam, including measurement of your vital signs.

At the end of every 2 cycles beginning with Cycle 4 (Cycles 4, 6, 8, and so on) blood (about 3-4 teaspoons) and urine will be collected for routine tests. You will have a CT or MRI.

If you are enrolled in the expansion group, blood (about 2 teaspoons each time) will be collected for PK testing before you take the daily dose of the study drug and then 1, 2, 4, 6, 8 and 24 hours later on Day 1 of Cycle 1. On Days 8, 15 and 21 of Cycle 1, blood (about 2 teaspoons each time) will also be collected for PK testing before you take the daily dose of the study drug and then 1, 2, 4, 6 and 8 hours later.

If you are enrolled in the expansion group, you will also have two mandatory tumor biopsies collected within 1- 7 days before you take your daily dose of the study drug and once during Days 15-21 of Cycle 1. To collect the biopsy, your doctor will insert a needle into the tumor and withdraw a small piece of the tumor. The tumor tissue will be studied to look at special "markers" in the tumor that may help researchers predict who may benefit from the study drug.

Length of Study:

You will remain on study until the disease gets worse, you decide to come off study, your doctor decides it is in your best interest to come off the study, you have intolerable side effects, or the sponsor closes the study.

If you decided to leave the study early you must tell the study doctor in writing and return any unused study drug. You must complete the end-of-study visit.

End-of-Study Visit:

Once you are off-study, you will have an end-of-study visit within 30 days after the last dose of PBI-05204. At this visit, the following tests and procedures will be performed:

* You will have a physical exam, including a measurement of your vital signs.
* You will have a performance status evaluation.
* You will have an ECG.
* You will have your heart rate monitored by a Holter monitor.
* Blood (about 3-4 teaspoons) and urine will be collected for routine tests
* You will have a CT/MRI scan to assess your tumors.
* Women who are able to have children must have a blood (about 2 teaspoons) or urine pregnancy test.

Long-Term Follow-up:

After you complete the end-of-study visit, your study doctor will continue to contact you or your family doctor for a minimum of 30 days. You may be contacted by a phone call (less than 5 minutes), and you will be asked about your general health.

This is an investigational study. PBI-05204 is not FDA approved or commercially available. At this time, PBI-05204 is only being used in research. Up to 52 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have an ECOG performance status score of 0-1
2. Histologic or cytologic diagnosis of a primary solid malignancy
3. Evidence (radiographic or tissue confirmation) that the disease is metastatic, or locally advanced in patients who are not candidates for standard therapy
4. Measurable disease, as defined by RECIST
5. Adequate bone marrow function defined as: a) absolute neutrophil count (neutrophil and bands) >/= 1,500 cells/mm3; b) platelet count >/= 100,000 cells/mm^3; c) hemoglobin >/= 9.0 g/dl
6. Adequate hepatic function defined as: a) total bilirubin </= 1.5 times the institutional upper limit ULN; b) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) </= 2.0 times the institutional ULN; c) Exception: patients with primary liver tumors or known liver metastases: </= 3.0 times the institutional ULN for AST and ALT
7. Adequate renal function defined as serum creatinine </= 1.5 times the institutional ULN
8. Serum potassium and magnesium levels within institutional normal limits. Total serum calcium or ionized calcium level must be greater than or equal to the lower limit of normal. Patients with low potassium, calcium and magnesium levels may be repleted to allow for protocol entry.
9. Prior chemo-, radio-, hormonal or immunotherapy are allowed. At least 4 weeks must have elapsed since the last chemotherapy or investigational agent (6 weeks for nitrosoureas, mitomycin-C, and liposomal doxorubicin), immunotherapy or radiotherapy and the beginning of protocol therapy. At least 2 weeks must have elapsed since last hormonal therapy or exposure to any other targeted kinase inhibitor (e.g., imatinib mesylate).
10. Men and women, ages 18 and older.
11. Women of childbearing potential (WOCBP) must be using an adequate method (i.e. barrier, spermicidal) of contraception to avoid pregnancy throughout the study and for a period of at least 1 month prior and at least 3 months after the study in such a manner that the risk of pregnancy is minimized.
12. continued from 11: WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea >/= 12 consecutive months; or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL].
13. continued from 12: Even women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential.
14. Participants must sign the written informed consent
15. Participants must be available for protocol-required follow-up

Exclusion Criteria:

1. WOCBP who are unwilling or unable to use an acceptable method (i.e. barrier, or spermicidal) to avoid pregnancy for the entire study period including the period from one month prior to starting study medication and for a period of at least 3 months after the study.
2. Women who are pregnant or breastfeeding.
3. Women with a positive pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) on enrollment or prior to study drug administration.
4. Men who are unwilling or unable to use an acceptable method (i.e. barrier, or spermicidal) of birth control for the entire study period and for at least 3 months after completion of study medication if their sexual partners are WOCBP.
5. Received extensive prior radiation therapy to the bone marrow. Generally, patients should have radiation to </= 25% of bone marrow-containing skeleton.
6. Symptomatic brain metastases that are either untreated or uncontrolled by surgery and or radiotherapy. Patients with symptoms of brain metastasis are not eligible unless brain metastasis are ruled out by CT or MRI and/or fully treated surgically or with WBRT.
7. A serious uncontrolled medical disorder or active infection which would impair the ability of the patient to receive protocol therapy.
8. Uncontrolled or significant cardiovascular disease, including: a) A myocardial infarction within 6 months b) Uncontrolled angina within 3 months c) Congestive heart failure within 3 months defined as NYHC-II d) Diagnosed or suspected congenital long QT syndrome
9. continued from 8: e) Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, Wolff-Parkinson-White (WPW) syndrome, or torsade de pointes). Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec). If the automated reading is prolonged (i.e., > 450 msec), the ECG should be manually overread. f) Any history of second or third degree heart block (may be eligible if currently have a pacemaker) g) Heart rate < 50 / minute on pre-entry electrocardiogram h) Uncontrolled hypertension (blood pressure >140 sys. and >90 dia.)
10. Dementia or altered mental status that would prohibit the understanding or rendering of informed consent
11. Patients who have not recovered from adverse events greater than grade 1 due to agents administered more than 4 weeks earlier.
12. Prior exposure to PBI-05204
13. Subjects taking these medications: digoxin/digitoxin, verapamil, amiodarone, propafenone, indomethacin, itraconazole, alprazolam, sotalol, and quinidine. Subjects taking non-potassium sparing diuretics (with the exception of lasix or furosemide) or other investigational drugs.
14. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.
15. Because patients with immune deficiency are at increased risk of lethal infections when treated with myelosuppressive therapy, patients known to have tested HIV-positive are excluded from the study.
16. Social situations that would limit compliance with study requirements.
17. History of allergic reactions attributed to compounds of similar chemical or biologic composition to PBI-05204, or other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Continuous assessment of safety throughout entire study period and determination of dose-limiting toxicities during and at the end of 28 Day Cycle(s).

CONTACTS AND LOCATIONS:
Overall Officials: David S. Hong, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Yang P, Menter DG, Cartwright C, Chan D, Dixon S, Suraokar M, Mendoza G, Llansa N, Newman RA. Oleandrin-mediated inhibition of human tumor cell proliferation: importance of Na,K-ATPase alpha subunits as drug targets. Mol Cancer Ther. 2009 Aug;8(8):2319-28. doi: 10.1158/1535-7163.MCT-08-1085. Epub 2009 Aug 11. PMID 19671733
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org